CLINICAL TRIAL: NCT06371365
Title: Prescription Pattern and Adverse Events of Postoperative Antithrombotic Regimes for Free Flap Surgery in Head and Neck Cancer
Brief Title: Adverse Events for Free Flap Surgery in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chi Lin, Director, Master Degree Program in Toxicology, Kaohsiung Medical University
Other Study IDs: KMUHIRB-E(II)-20220204
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Surgical Flaps; Flap Failure Risk Factors; Hematoma Risk Factors; Thrombosis Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent free flap surgery
  Interventions: Procedure: Free Flap surgery

INTERVENTIONS:
Procedure: Free Flap surgery — No intervention, this is an observational study

SUMMARY:
This is a cohort study collecting patients with head and neck cancer who underwent free flap surgery at a single medical center between January 2019 and January 2022.

DETAILED DESCRIPTION:
Patient information are collected from the electronic medical records retrospectively:

Head and Neck cancer diagnosis: The International Classification of Diseases, Tenth Revision (ICD-10), which included C00-C14, C31, C32, C73, C75.0, C75.4 and C41.1.

The cancer stage, alcohol use, betel nut, and smoking, and baseline comorbidities.

Surgical characteristics including flap history, ablation time, reconstruction time, donor sites, recipient sites, neck dissection, flap size, anastomosis, artery types, vein types, intraoperative sealants used, and intravenous calcium channel blocker nicardipine to control hypertension after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater and equal to 20 years old
* Underwent free flap surgery
* Had head and neck cancer

Exclusion Criteria:

* HIV positive
* Pregnant, breast feeing women
* Missing surgical charts

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient greater than or equal to 20 years old who had free flap surgery following cancer ablation for head and neck cancer.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with flap failure | 30 days post-operation
  Flap necrosis with a need for a new flap or other surgical procedures.

SECONDARY OUTCOMES:
Number of participants with hematoma | 30 days post-operation
  Surgical indication for reoperation. Reoperation is performed when patients experienced major complications refractory to bedside management.
Number of participants with thrombosis | 30 days post-operation
  Surgical indication for reoperation. Reoperation is performed when patients experienced major complications refractory to bedside management.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chi Lin, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsiung PH, Huang HY, Chen WY, Kuo YR, Lin YC. Cumulative risk factors for flap failure, thrombosis, and hematoma in free flap reconstruction for head and neck cancer: a retrospective nested case-control study. Int J Surg. 2024 Dec 1;110(12):7616-7623. doi: 10.1097/JS9.0000000000002069. PMID 39236088